CLINICAL TRIAL: NCT02015598
Title: Comparison of Oral Intake of Antioxidant Carbocysteine and Nasal Continuous Positive Airway Pressure (CPAP) for Treating in Moderate and Severe Obstructive Sleep Apnoea Syndrome Patients : a Randomized Clinical Trial
Brief Title: Antioxidant Carbocysteine Treatment in Obstructive Sleep Apnoea Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Kang Wu, master, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRD201319
Record Dates: First submitted 2013-12-10; First posted 2013-12-19 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Obstructive Sleep Apnoea
Keywords: Obstructive sleep apnoea; Antioxidant; drug treatment; oxidative stress; Continuous Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Carbocysteine; Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbocysteine (Experimental): Carbocysteine , tablet ,250mg per one tablet , patients oral intake with 500mg .tid.(1500mg/day)
  Interventions: Drug: Carbocysteine
- Continuous Positive Airway Pressure (Active Comparator): Continuous Positive Airway Pressure(CPAP),auto-CPAP(USA,Philips), patients use Nasal CPAP overnight.
  Interventions: Device: Continuous Positive Airway Pressure

INTERVENTIONS:
Drug: Carbocysteine — carbocisteine (2×250 mg, three times daily) for 6 weeks. The tablets are provided by Baiyunshan Pharmaceutical, China. patients will interviewed after 3 weeks to check their adherence to the study regimen by collecting and counting the number of remaining tablets, record adverse events, and refill study tablets for the next 3 weeks.
  Other Names: S-Carboxymethylcysteine; SCMC
  Arms: Carbocysteine
Device: Continuous Positive Airway Pressure — Patients will interviewed after 3 weeks and the end of trial.We will check their compliance to device memory download , record adverse events and pressure .
  Other Names: Nasal Continuous Positive Airway Pressure
  Arms: Continuous Positive Airway Pressure

SUMMARY:
Obstructive sleep apnoea syndrome (OSAS) is characterised by repeated episodes of upper airway occlusion during sleep.It can cause cycles of hypoxia reoxygenation. And it was postulated that intermittent hypoxia seems to resemble ischemia-reperfusion.Many study suggest that ischemia-reperfusion represents an oxidative stress causing increased generation of reactive oxygen species, especially superoxide anions.It is one of the most important mechanisms of cardiovascular diseases, including hypertension, coronary artery disease and cerebrovascular accident complication with OSAS.So many individuals approve OSAS is an Oxidative Stress disease.

Continuous positive airway pressure (CPAP) is the first-line of treatment method in moderate/severe OSA.But poor adherence to CPAP treatment is very common.The failure rate with CPAP treatment is more than 50%.So we are searching a new treatment for that patients. Carbocysteine is a antioxidant.It can not only scavenges the free radicals but also replenishes glutathione(GSH)which is has double antioxidant capacity. However, Carbocysteine is cheaper than other which has double antioxidant capacity drugs,such as N-acetylcysteine.The purpose is to evaluate efficacy of oral intake of Antioxidant Carbocysteine witch can reduce oxidative stress and improve the symptom of OSAS.It recover the imbalance in the oxidant-anti-oxidant status may reduce cardiovascular abnormalities in Patients with OSAS.

DETAILED DESCRIPTION:
OSAS patients are required to fill in questionnaire.And Inflammation biomarkers and Oxidative Stress biomarkers and ultrasonic will be tested.Then patients are randomly allocated to one of two groups. One group is treated with oral intake of Antioxidant Carbocysteine 500mg tid. The second group is treated with CPAP. After 6 weeks treatment, all patients will take the overnight polysomnogram test again, and take questionnaire, blood , ultrasonic test.

ELIGIBILITY:
Inclusion Criteria:

1. Male in an age range of 18 to 65 years
2. Obstructive Sleep Apnoea with an Apnea Hypopnea Index (AHI) of greater than or equal to 15 confirmed by polysomnography
3. The patient is able to provide consent
4. The patient were not receiving therapy for sleep apnoea,such CPAP or surgery.

Exclusion Criteria:

1. Inability to tolerate Carbocysteine or CPAP
2. Treatment with CPAP or surgery prior to or at the time of enrolment
3. presence of active acute or chronic infection
4. Patients with unstable cardiovascular diseases (unstable angina, myocardial infarction, stroke, or transient ischemic attacks), neuromuscular diseases, chronic respiratory diseases, peripheral vascular disease
5. Using of steroidal , nonsteroidal anti-inflammatory, vasodilators ,lipid-lowering drugs,or other medications that lower oxidative stress.
6. Intake of central relevant drugs, sedatives, or other drugs which impair sleep
7. Unwilling to participate in the study
8. Participation in another clinical study in the past 4 weeks
9. Shift worker

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change of polysomnography (PSG) parameters after oral intake of Carbocysteine treatment | after 6 weeks
  The Carbocysteine group will oral intake of Carbocysteine 500mg,tid for 6 weeks.We will examine the compliance with the drugs by Recycling the rest of the tablets.We compare the improvement of PSG parameters,such as AHI ,oxygen desaturation index(ODI),oxyhemoglobin saturation.
Daytime sleepiness(EDS) after oral intake of Carbocysteine treatment | after 6 weeks
  EDS is evaluated by Epworth Sleeping Scale(ESS) grade.ESS≥9 means EDS.The higher the ESS, the more daytime sleepiness they feel.
Change of Oxidative Stress after oral intake of Carbocysteine treatment | after 6 weeks
  Biomarkers is measured from venous blood.The blood is collected in the morning .After centrifugation ,the supernatant was kept at -80 degree centigrade.

SECONDARY OUTCOMES:
Evaluate efficacy of oral intake of Antioxidant Carbocysteine in comparison to Nasal continuous positive airway pressure (CPAP) treatment . | after 6 weeks treatment
  We will examine the compliance with CPAP device memory download.We will compare the two group by the PSG parameters ,ESS, and Biomarkers .

OTHER OUTCOMES:
Change of vascular function after oral intake of Antioxidant Carbocysteine | after 6 weeks after oral intake of Carbocysteine treatment
  Vasoreactivity Testing Protocol and intima-media thickness is measured by high-resolution ultrasonography at baseline and 6 weeks after treatment.Vasoactive mediators from blood will be studied.

CONTACTS AND LOCATIONS:
Overall Officials: NuoFu Zhang, professor, Principal Investigator — Guangzhou Institute of Respiratory Disease
Locations (1):
- Guangzhou institute of respiratory disease, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Wu K, Su X, Li G, Zhang N. Antioxidant Carbocysteine Treatment in Obstructive Sleep Apnea Syndrome: A Randomized Clinical Trial. PLoS One. 2016 Feb 5;11(2):e0148519. doi: 10.1371/journal.pone.0148519. eCollection 2016. PMID 26849119